CLINICAL TRIAL: NCT02742675
Title: OMPCa-Shanghai: An Open-label, Randomized Prospective Phase II Trial of Androgen Deprivation Therapy or Androgen Deprivation Therapy Plus Definitive Treatment (Radiation or Surgery) of the Primary Tumor in Oligometastatic Prostate Cancer
Brief Title: Androgen Deprivation Therapy or Androgen Deprivation Therapy Plus Definitive Treatment (Radiation or Surgery)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-OMPCa
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; androgen deprivation therapy; local treatment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; Flutamide; Leuprolide; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- androgen deprivation therapy (Experimental): Patients will receive androgen-deprivation therapy comprising luteinizing-hormone releasing-hormone (LHRH) agonist (leuprolide acetate, goserelin acetate, buserelin, or triptorelin) subcutaneously or as an injection AND an oral antiandrogen therapy (flutamide 3 times daily or bicalutamide once daily).
  Interventions: Drug: Bicalutamide; Drug: goserelin acetate; Drug: flutamide; Drug: leuprolide acetate; Drug: triptorelin
- androgen deprivation therapy plus definitive treatment (Experimental): Patients will receive androgen-deprivation therapy as in arm I in addition to definitive treatment including surgery to remove prostate or radiation therapy to the prostate.
  Interventions: Drug: Bicalutamide; Drug: goserelin acetate; Drug: flutamide; Drug: leuprolide acetate; Drug: triptorelin; Procedure: Definitive Treatment

INTERVENTIONS:
Drug: Bicalutamide — Given orally
  Other Names: Casodex
Drug: goserelin acetate — Given subcutaneously or as an injection
  Other Names: Zoladex
Drug: flutamide — Given orally
  Other Names: Eulexin
Drug: leuprolide acetate — Given subcutaneously or as an injection
  Other Names: Enantone
Drug: triptorelin — Given subcutaneously or as an injection
  Other Names: Diphereline
Procedure: Definitive Treatment — surgery to remove prostate or radiation therapy to the prostate.
  Arms: androgen deprivation therapy plus definitive treatment

SUMMARY:
The goal of this clinical research is to learn if treatment with androgen deprivation therapy in combination with surgery or radiation therapy can prolong the progression-free survival of oligometastatic prostate cancer than androgen deprivation therapy alone. The safety of this treatment combination will also be studied.

DETAILED DESCRIPTION:
Today androgen deprivation therapy has been a standard treatment for metastatic prostate cancer, but as to the special type of prostate cancer-oligometastatic prostate cancer, except for androgen deprivation therapy, whether local treatment can be the part of treatment for it? The purpose of this study is to evaluate whether local treatment combined with androgen deprivation therapy can extend progression-free survival, as well as overall survival and life quality of patients of oligometastatic prostate cancer compared with androgen deprivation therapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients;
2. 18 yrs and older, and 80 yrs and younger;
3. Histologically or cytologically proven prostate carcinoma;
4. Documented evidence of M1 disease by AJCC (American Joint Committee on Cancer) staging by Bone scan, CT and/or MRI; and metastatic lesions are limited to the lymph nodes or bones, at the same time the number of lesions should less than or equal to 5;
5. ECOG PS 0 or 1;
6. Treatment initiation with androgen deprivation therapy no longer than 6 months prior to randomization;
7. Life-expectancy based on comorbid conditions >2 years;
8. No serious medical complications;
9. The primary lesion of prostate cancer has not yet received local treatment;
10. Must be a candidate for surgery and/or radiation therapy and follow-up and the treatment will not bring about serious complications to patients;
11. Ability to understand and willingness to sign informed consent.

Exclusion Criteria:

1. Had received treatment for primary lesion, including: radical prostatectomy, radical radiation therapy and so on;
2. Patients who received systemic chemotherapy before;
3. Androgen deprivation therapy time is greater than six months;
4. Visceral organ metastasis (liver, lung, brain and other organs);
5. Small cell carcinoma of the prostate;
6. Psychiatric or medical conditions which, in the opinion of the treating physician, would not allow the patient to undergo the proposed treatments safely;
7. Patients who are not willing to accept the complications caused by the treatment to primary lesion;
8. Combined with other malignant tumor history (in addition to the skin basal cell carcinoma or other tumors that have been cured more than five years);
9. Other serious diseases, for example: unstable heart disease after treatment, myocardial infarction in 6 months prior to treatment, cardiac function grade 3-4 (NYHA); high blood pressure that can not be controlled after medical treatment (greater than 150/90mmHg); serious neurological or mental disorders, including dementia and epilepsy; uncontrolled active infection; acute gastric ulcer; hypocalcemia; chronic obstructive pulmonary disease that needs hospital treatment;
10. Has participated in other clinical research before.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (radiographic progression-free survival) | 2 years

SECONDARY OUTCOMES:
Overall survival | 3 years
time of PSA progression | 3 years
the quality of life | 3 years
  Quality of Life assessed by the EORTC QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ye Dingwei, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dai B, Zhang S, Wan FN, Wang HK, Zhang JY, Wang QF, Kong YY, Ma XJ, Mo M, Zhu Y, Qin XJ, Lin GW, Ye DW. Combination of Androgen Deprivation Therapy with Radical Local Therapy Versus Androgen Deprivation Therapy Alone for Newly Diagnosed Oligometastatic Prostate Cancer: A Phase II Randomized Controlled Trial. Eur Urol Oncol. 2022 Oct;5(5):519-525. doi: 10.1016/j.euo.2022.06.001. Epub 2022 Jun 29. PMID 35780048